CLINICAL TRIAL: NCT06590025
Title: A Phase III, Randomized, Active Comparator-controlled, Clinical Trial to Study the Efficacy and Safety of the INtegral Cognitive REMediation Program (INCREM) in Patients with Depression
Brief Title: Study the Efficacy and Safety of the INtegral Cognitive REMediation Program (INCREM) for Depression
Acronym: INCREM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-RID-2022-125
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Depression; Depressive Disorder
Keywords: cognitive symptoms; cognitive remediation; rehabilitation; major depressive disorder; functional recovery
MeSH Terms: conditions — Depression; Depressive Disorder; Neurobehavioral Manifestations; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is randomized clinical trial comparing two psychological interventions: INCREM and psychoeducation, and no drugs or biological/vaccine or combination products are tested, regardless it is a phase 3 study. Included patients can be prescribed pharmacological treatments, but these are not investigated here-in.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INtegral Cognitive REMediation program (INCREM) (Experimental): The functional remediation (FR) program of INCREM intervention consists of 12 sessions (1s/wk) in a group format, which is devoted to improve the daily functioning of patients and therefore, is based on very ecological tasks where compensation techniques are used. An computerized cognitive training will follow the INCREM arm in individual sessions. 12 individually tailored modules of 20 minutes will be created with a licensed software (NeuronUp).
  Interventions: Behavioral: INtegral Cognitive REMediation program
- PSYCHOEDUCATION (Active Comparator): The psychoeducation program for Major Depression was also developed in the context of the previous project (PI17/00056). It consists of 12 sessions (1s/wk) in a group format and includes all aspects related to MDD (Raventós, González & Portella. Protocolo de Psicoeducación para depresión. Ed Permanyer: Barcelona. 2020). To ensure the similarity between the two intervention arms, in the comparator arm, participants will play a previously selected mental skill game on a digital device for 20 minutes.
  Interventions: Behavioral: Psychoeducation for depression

INTERVENTIONS:
Behavioral: INtegral Cognitive REMediation program — This comprehensive functional remediation program includes a traditional CR component with a specialized therapist (based on the compensation model) and a CCT component adapted to the difficulties of each patient. The inclusion of both aspects allows adapting the intervention to the present difficulties by forming new strategies with compensation techniques and promoting translation to everyday life. Therefore, the intervention aims at improving cognitive functioning (beyond a mere training) so as to facilitate the improvement and maintenance of psychosocial functioning for patients with MDD.
  Other Names: INCREM
  Arms: INtegral Cognitive REMediation program (INCREM)
Behavioral: Psychoeducation for depression — Psycho-education refers to educating individuals about depression and the various treatment options. It is a form of therapy that aims to provide individuals with the knowledge and skills to manage their mental health symptoms effectively.
  Arms: PSYCHOEDUCATION

SUMMARY:
Feeling sad about negative or stressful events has nothing to do with the diagnosis of depression, as this is a very prevalent mental illness among the population with devastating consequences for the person suffering from it. Symptoms range from mood swings, extreme sadness, apathy, inability to feel pleasure, to sleep problems, eating disorders, physical problems, and more. Other very common but little-known symptoms are those that affect memory, concentration, and the ability to organize and solve problems.

Recent scientific findings have shown that these symptoms, called cognitive symptoms, are the most interfering with day-to-day life, even when other mental symptoms begin to improve or have resolved. Cognitive symptoms are associated with work difficulties, especially in terms of productivity or a decrease in social relationships to the point of isolation, thus interfering with the full recovery from depression. Studies have estimated that the economic and social costs not related to the health costs of depression can be more than 90 million euros per year. The fact that cognitive symptoms are not explored during clinical interviews means that they are not treated adequately, and professionals usually wait for cognitive difficulties to be resolved with the available antidepressant treatments. But more than 30% of people with depression are unable to return to work, and up to 45% of patients are on sick leave a year later, although mood symptoms have often been ameliorated.

This opens a new line of research worldwide that aims to find effective treatments for the cognitive symptoms of depression. Some drugs have been developed and cognitive training programs designed for patients with dementia or neurological conditions have been tested, but the results are not convincing enough because there is no transfer of cognitive improvements into people&amp;amp;#39;s lives. The research team of this proposal designed a comprehensive rehabilitation program for cognition and daily functioning for depression, taking into account the specific cognitive symptoms, and the real difficulties that patients face. Thus was born INCREM (INtegral Cognitive REMediation for Depression), which includes cognitive training and therapy sessions focused on the rehabilitation of daily functioning. The first results in very selected samples have shown an objective improvement in day-to-day functioning, not only after the intervention but up to 6 months later. The aim of this proposal is to demonstrate the effectiveness and benefits of INCREM for depression in a larger and more diverse sample of patients, as well as finding out the effects of INCREM on the brain. The ultimate goal is to implement this type of therapy in mental health care centers in order to treat patients&amp;amp;#39; cognitive symptoms and get them back to their personal, work and social lives.

DETAILED DESCRIPTION:
BACKGROUND: Major Depressive Disorder (MDD) is a mood disorder that places substantial clinical, social and economic burden onpatients, as well as on their families and wider society. The total cost of MDD is estimated at 170,000 million euros per year (www.euro.who.int), where more than a half are indirect costs such as loss of productivity in the workplace, sick leave and early retirement. In Spain, it is estimated that depression causes complete functional disability of 47 days per year on average and partial functional disability of 60 days per year (1). Particularly in Catalonia, depression had a direct health cost of €155 million, which rose to €735 million when lost productivity was included (temporary disability: 27%; permanent: 48%) in the last decade (2). The authors concluded that the cost of mental illness has a considerable impact from asocietal perspective, as direct costs in the public health system or indirect costs related to productivity losses are only part of total costs of depression (3). Some studies confirm that severity of depressive symptoms predicts the functional deterioration of patients, beyond losing a job or spending public health resources. More recent studies add that cognitive symptoms (i.e., alterations in executive functions, attention, memory and processing speed) are even more important independent predictors of such psychosocial dysfunction in subsequent depressive episodes (4). Therefore, cognitive symptoms could explain the low full recovery rates and the functional disability of patients with MDD (5,6). Although cognitive symptoms are nowadays recognized and partially incorporated as a criterion for the diagnosis of an episode of MDD (DSM-5), until recently no treatment addressed these symptoms. There is increasing evidence that patients with MDD show heterogeneity in cognitive difficulties, presenting different cognitive profiles in the first depressive episode as demonstrated in project PI13/01057 (IP: Maria J Portella) and in the different stages of the disease (7). Up to 45% of patients with treated MDD have permanent cognitive deficits (8), which significantly interfere with work and daily functioning (9).

Some evidence has acknowledged the poor efficacy of most pharmacological treatments in the improvement of cognitive symptoms (10). Although new antidepressants with other mechanisms of action seem to have different effects on the cognitive function, these still show low or moderate efficacy. Regarding non-pharmacological treatments, cognitive remediation (CR) has been investigated as a possible treatment of cognitive dysfunction of depressive disorders in the last decade. But the results are not fully satisfactory and efficacy is in its infancy. Different reasons have been suggested to explain the low impact of cognitive rehabilitation programs for MDD, among which the use of neurological models in the design of these programs, instead of using compensatory techniques more effective in psychiatric disorders (11); or the fact of not taking into account the episodic nature and tendency to chronicity of MDD, which implies very different profiles of cognitive involvement among patients (7). Therefore, a critical aspect of remediation programs for MDD is to adapt them to the cognitive profile of each patient.

In an attempt to improve previous results using poorly structured programs, computerized cognitive training (CCT) had proven to be more beneficial than available CR programs in patients with MDD (12). This type of training was based on mental tasks repetition, which ended up having an effect on patients' difficulties. Subsequently, several studies have shown that CCT is perhaps the best method of administration for MDD, as tasks are adjusted to the needs of each individual. In a meta-analysis including the 9 randomized studies that existed of CCT in MDD (13) it was observed how CCT was associated with a slight improvement of depressive symptoms but scarcely of daily functioning. In this regard, it should be noted that only two of the nine studies investigated the impact of treatment on global functioning specifically. Regarding cognitive benefits, the results depended on cognitive domains, seeing a notable improvement in working memory and attention, while executive functions and verbal memory remained altered. These benefits were not easily transferred to new tasks or only when they required the same processing requirements as trained tasks. Thus, one of the biggest problems of these computerized programs was the transfer of trained skills to daily life tasks, including work capacity. Another recent approach is the Goal Management Training (GMT), a strategy-based CR intervention. The findings comparing GMT with drill-and-practice CCT has shown long-term mental health following GMT, while improvements in everyday life might require additional treatment or maintenance to sustain (14). Sample sizes of previous works are extremely limited (n&amp;lt;30), casting doubt on the representativeness of findings and thus impeding their generalization or implementation to real-world clinical settings. The study on Functional Remediation (FR) with the largest sample was carried out by the group of Martínez-Aran for patients with bipolar disorders in a multicentre clinical trial which showed efficacy of FR compared to treatment as usual (TAU) or psychosocial functioning (15). However, these programs did not include any tailored cognitive intervention at the individual level, such as CCT, and therefore the transfer of cognitive improvement to daily functioning was not achieved.

The mechanism of action of cognitive remediation interventions is still unknown. Very few studies have investigated biomarkers associated to CR response, apart from a unique study (11). There is mounting evidence that neurotrophic factors, immune markers and oxidative stress play a key role in cognitive dysfunction (16-20), regardless of underlying psychiatric pathology. Research of peripheral biomarkers and treatment response have described fairly consistent findings, in which neuroimmune alterations back to normal levels (16,17). Magnetic resonance imaging (MRI) evidence suggests a possible link between structural/functional anomalies in the brain and on one hand, a decrease of growth factors and on the other, an increase of circulating inflammation and oxidative markers. Several of these studies have been carried out by the PI, as well as other members of the consortium (see references). Mostly, neuroimaging studies have reported alterations in brain regions involving fronto-temporal and cortico-limbic circuits (21), also related with pharmacological treatment response and prediction of recurrence (22) in the areas mentioned above, where smaller brain volumes typically estimate poorer treatment response, whereas larger brain volumes correlate with good response and remission. Less consensus has been achieved with white matter alterations (investigated with diffusion tensor imaging (DTI), where some studies report lower white matter fractional anisotropy (FA) in good response to treatment, while others show the opposite (23). Other inconsistencies are found in functional MRI (fMRI) in treatment response, especially in task-based fMRI, but also in resting-state functional connectivity (RSFC), partially due to a considerable variability in study designs (24). One of the recent MRI technical advances is to study microstructural changes in both grey and white matter, more expectable to be detected in usually normal-appearing brains (i.e., without atrophy o severe /detectable white matter hyperintensities). One limitation of previous studies was the application of gross neuroimaging techniques that may not capture subtle cortical changes driving cognitive and behavioural outcomes. DTI has now been proposed to measure both cortical (grey matter) and subcortical (white matter) changes using mean diffusivity (MD) metrics, overcoming former technical difficulties for the study of cortical microstructure. Cortical MD is a measure of cortical microstructure integrity and has proven to be a sensitive tool for subtle cortical changes in early stages of neurodegenerative diseases (24).

However, most of the randomized controlled trials of CR or CCT effects in psychiatric and neurologic conditions use clinical endpoints that may be soaked in subjectivity, or surrogate endpoints based on psychometric tools. Blood and neuroimaging biomarkers may therefore represent a clinically applicable alternative surrogate endpoints that would be cost-effective and minimally invasive so as to provide the neurobiological underpinnings of functional and cognitive remediation response.

STATE-OF-THE-ART: Based on the evidence of unfavourable findings, in 2017 a project was granted for the development of INtegral Cognitive REMediation for Major Depression (INCREM), (PI17/00056, IP: Maria J Portella). This comprehensive functional remediation program includes a traditional CR component with a specialized therapist (based on the compensation model) and a CCT component adapted to the difficulties of each patient. The inclusion of both aspects allows adapting the intervention to the present difficulties by forming new strategies with compensation techniques and promoting translation to everyday life. Therefore, the intervention aims at improving cognitive functioning (beyond a mere training) so as to facilitate the improvement and maintenance of psychosocial functioning for patients with MDD. The details of INCREM program have been published as a protocol (25).

The proof-of-concept revealed very promising findings. Preliminary data was acquired through a randomized clinical trial, which included 3 treatment arms: INCREM (active arm), a psychoeducation program (active comparator arm) and usual treatment (TAU, non-active arm). Such a change in the methodology made it impossible to demonstrate the efficacy of the program, but the pilot study has served to demonstrate the feasibility of INCREM. The results showed that INCREM significantly improved psychosocial functioning in remitted depressed patients soon after the end of the intervention and six months after (26). More than 65% of patients achieved functional recovery. There was also an enhancement of general cognition, providing evidence of the necessity to combine compensatory and drill-and-practice strategies. The acceptability of the interventions (explored through open question to all participants) varies from good to very good. More importantly, this previous study demonstrates the feasibility, safety and benefits of INCREM. The efficacy of the INCREM program with respect to the psychoeducation intervention is now being analysed through a multicentre randomized clinical trial, which was funded by the ISCIII call (PI20/00270, IP: Maria J Portella) and covers different sociodemographic areas. Preliminary findings point towards the confirmation of significant improvement of long-term psychosocial functioning, as well as enhancement of cognitive functioning and of overall patients' well-being. The inclusion of comprehensive data, other than clinical outcomes, should be part of future studies. The integration of clinical, neuroimmuno-oxidative factors and fine neuroimaging markers will improve the study of INCREM outcomes, and therefore, the accuracy and sensitivity of the prediction for this particular treatment response.

The present call offers an exceptional opportunity to continue this innovative and promising line of research started by the PI, in which most of the members of the research team have been involved. This Phase III clinical trial will involve a much larger group of patients and will focus on determining whether INCREM would be safe and effective for a wide variety of patients with depressive disorders. This should confirm and expand the efficacy of INCREM, and more importantly, should help depressed patients with cognitive symptoms achieving full recovery, which in turn should represent significant decrements of public health and social-personal costs associated to depression.

HYPOTHESES

1. Patients in the INCREM arm will improve their functional and cognitive functioning, showing:

   * an improvement in psychosocial functioning on the FAST scale (main variable)
   * a mid-term improvement in pragmatic psychosocial variables: reduction in the number of sick leaves, increment of self efficacy measures related with work and social activities.
   * an improvement in cognitive performance both in objective cognitive tests and subjective appraisal.
2. Patients in the INCREM arm will achieve full recovery (i.e., global clinical, functional and cognitive symptoms amelioration).
3. INCREM will reduce the number of relapses and improve subsyndromic symptoms.
4. functioning and cognitive improvements will be associated with neuroimmune-oxidative markers. Specifically:

   * increments of neurotrophic markers will be associated with decrements of psychosocial and cognitive dysfunction
   * decrements of oxidative stress markers will be associated with decrements of psychosocial and cognitive dysfunction
   * decrements of pro-inflammatory markers will be associated with decrements of psychosocial and cognitive dysfunction
   * microstructural grey and white matter changes will be associated with percentage change in psychosocial and cognitive scales.

OBJECTIVES Main

1. To demonstrate the efficacy of INCREM program through a randomized clinical trial with an active comparator (psychoeducation) in a representative sample of patients with depressive disorders.
2. To improve the global functioning (through aiming full recovery) of patients with depressive disorders.
3. To determine the mechanism of action on INCREM by using neurobiological biomarkers that may serve as surrogate clinical endpoints of the efficacy of INCREM.

Secondary

1. To use individual cognitive profiles of patients with MDD to personalize the content of CCT so as to achieve full recovery.
2. To increase the effect size of the results of INCREM with respect to previous phases, which were run in limited samples:

   * by using a larger sample, from different geographical settings and in a wider spectrum of depression.
   * by including compensatory and drill-and-practice strategies.
   * by combining traditional groups sessions + individualized cognitive training.
3. To study the specific clinical, sociodemographic factors (i.e., psychosocial and self-efficacy) and biomarkers that mediate the potential clinical and functional improvement.

STUDY DESIGN Randomized, multicentre, blind evaluator, controlled with active comparator clinical trial (Phase III), stratified by biological sex, age, and level of studies to assess the efficacy of the INCREM program (functional rehabilitation and computerized cognitive training). The main variable will be the improvement in global psychosocial functioning -average change in the FAST (Functioning Assessment Short Test) score between baseline (T0), post-treatment (T1) and follow-up (6 mo after the end of intervention; T2).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 y.o. and beyond with a remitted or active episode of major depression (DSM-5 criteria; maximum score of 18-20 on the HDRS-17)
* showing cognitive symptoms (scores below 80 on the SCIP)
* with functional difficulties (scores above 12 on the FAST).

Exclusion Criteria:

* IQ below 85;
* any unstable or inadequately-treated medical condition that may affect neuropsychological performance;
* being under drug treatment in the last 4 weeks with glucocorticoids, probiotics, non-steroidal anti-inflammatory drugs, bile acid sequestrants, immunosuppressive drugs, anti-histamines, mast cell stabilizers, and antioxidant supplements;
* use of systemic antibiotics the last 2 months;
* presence of any comorbid psychiatric condition, other than personality disorders or nicotine use disorders, in the last three months;
* for bipolar disorders, presence of a manic or mixed episodes in the last three months;
* accomplish criteria for severe treatment resistant depression;
* patients who had received electroconvulsive therapy in the previous year;
* patients receiving any other structured psychological intervention in the 3 months prior to the study;
* not having the necessary electronic means (computer or tablet) or internet connection to be able to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological sex assigned at birth (female, male, non-binary)
Enrollment: 296 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functioning Assessment Short Test (FAST) | From enrollment to the end of treatment (12 weeks) and to the end of follow-up (6 months)
  The FAST is a valid, widely used instrument to test psychosocial functioning. The main outcome measure will be the percentage of change in FAST scores between T0 and T1 and T2.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale-17 items (HDRS_17) | From enrollment to the end of treatment (12 weeks) and to the end of follow-up (6 months)
  This scale iss used to rate the severity of depression symptoms by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms.
Remission from Depression Questionnaire (RDQ) | From enrollment to the end of treatment (12 weeks) and to the end of the follow-up (6 months)
  The RDQ is a reliable and valid measure that evaluates the multiple domains that depressed patients consider important in determining remission.
Screening for Cognitive Impairment in Psychiatry (SCIP) | From enrollment to the end of the intervention (12 weeks) and to the end of the follow-up (6 months)
  The SCIP is a brief and easy-to-administer tool, requiring the test sheet, a clock and a pencil only, specifically targeting psychiatric populations.
Perceived Deficits Questionnaire for Depression (PDQ-R) | From enrollment to the end of the intervention (12 weeks) and to the end of follow-up (6 months)
  The PDQ-D is a self-reported scale for monitoring cognitive dysfunction in patients with major depression. The PDQ-D is a modified version of the original PDQ, which was developed to assess cognitive symptoms in patients with multiple sclerosis.
Functional and structural brain changes (magnetic resonance imaging) | From enrollment to the end of follow-up at 6 months
  Two functional and structural scans will be obtained of each individual (randomly selected subsample; n=40) to determine the potential mechanism of action of INCREM

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Portella, Dr, Principal Investigator — Institut de Recerca Sant Pau
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
There may be competitive interests involved, particularly if the data could provide an advantage to other researchers, but we do not rule out in future. In any case, because the data sharing policies and regulations of the institution may restrict the dissemination of such information, the potential share of data has been included in the informed consent sheet for participants.